CLINICAL TRIAL: NCT05708235
Title: A Proof of Concept Study to Evaluate Treatments' Efficacy by Monitoring Minimal Residual Disease Using ctDNA in HR-positive/HER2-negative Early Breast Cancer Population
Brief Title: A PoC Study to Evaluate Treatments' Efficacy by Monitoring MRD Using ctDNA in HR-positive/HER2-negative EBC Population
Acronym: MiRaDoR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MedSIR (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MedOPP485
Record Dates: First submitted 2023-01-12; First posted 2023-02-01 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — giredestrant; abemaciclib; inavolisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm A: Control Arm (No Intervention): Patients must continue the same standard ET,prescribed as per standard practice, used in the surveillance phase. Changes in ET are not allowed.
- Arm B: Experimental Arm with giredestrant (Experimental): Giredestrant: 30 mg will be taken orally (PO) once a day (QD) on Days 1 to 28 of each 28-day cycle up to five years or until disease recurrence, unacceptable toxicity, or treatment/study discontinuation (whichever occurs first).
  Interventions: Drug: Giredestrant
- Arm C: Experimental Arm with giredestrant + abemaciclib (Experimental): * Giredestrant: 30 mg will be taken PO QD on Days 1to 28 of each 28-day cycle up to five years or until disease recurrence, unacceptable toxicity, or treatment/study discontinuation (whichever occurs first).
  * Abemaciclib 150mg will be taken PO twice daily (BID) (two intakes for a total daily dose of 300 mg) during each 28-day cycle up to two years or until disease recurrence, unacceptable toxicity, or treatment/study discontinuation (whichever occurs first).
  Interventions: Drug: Giredestrant; Drug: Abemaciclib
- Arm D: Experimental Arm with giredestrant + inavolisib (Experimental): * Giredestrant: 30 mg will be administered PO QD on Days 1-28 of each 28-day cycle up to five years or until disease recurrence, unacceptable toxicity, or treatment/study discontinuation (whichever occurs first).
  * Inavolisib: 9 mg will be administered PO QD on Days 1-28 of each 28-day cycle up to two years or until disease recurrence, unacceptable toxicity, or treatment/study discontinuation (whichever occurs first).
  Interventions: Drug: Giredestrant; Drug: Inavolisib

INTERVENTIONS:
Drug: Giredestrant — Giredestrant is a highly potent, non-steroidal, oral selective ER antagonist and degrader (SERD)
  Other Names: GDC-9545
  Arms: Arm B: Experimental Arm with giredestrant; Arm C: Experimental Arm with giredestrant + abemaciclib; Arm D: Experimental Arm with giredestrant + inavolisib
Drug: Abemaciclib — Abemaciclib is an orally administered CDK4/6 inhibitor
  Other Names: LY2835219
  Arms: Arm C: Experimental Arm with giredestrant + abemaciclib
Drug: Inavolisib — Inavolisib is a potent, selective inhibitor of the Class I phosphatidylinositol 3-kinase α (PI3K-alpha isoform (p110-alpha)
  Other Names: GDC-0077
  Arms: Arm D: Experimental Arm with giredestrant + inavolisib

SUMMARY:
This trial is a multicenter, open-label, non-comparative, phase II, biomarker-driven adjuvant treatment study involving the periodic collection and analysis of blood samples from patients with HR-positive/HER2-negative early-stage BC at higher risk of relapse, who have undergone surgery within the previous five years, with no evidence of locoregional, contralateral, or distant disease.

The study design is composed by an initial pre-screening phase, a molecular follow-up phase (ctDNA surveillance phase), and an interventional therapeutic phase (treatment phase).

After informed consent is obtained, a total of1,260 eligible patients will enter a ctDNA surveillance in which primary tumor tissue and matched normal blood will be collected from each patient to obtain a patient-specific somatic mutations panel (tumor signature).

At the event of ctDNA positivity, patients will be screened to enter the treatment phase of the study. Upon confirmed eligibility, a total of 40 patients will be allocated in one of the following trial's arms adopting a sequential recruitment strategy:

Arm A: Control Arm (N=10) Arm B: Experimental Arm with giredestrant (N=10) Arm C: Experimental Arm with giredestrant + abemaciclib (N=10) Arm D: Experimental Arm with giredestrant + inavolisib (N=10)

If the strategy of ctDNA monitoring enables physicians to identify patients at high risk of relapse and assess whether treatment at molecular relapse can improve outcome, new cohorts may be added to the study.

DETAILED DESCRIPTION:
This is a multicenter, open-label, non-comparative, phase II, biomarker-driven adjuvant treatment study involving the periodic collection and analysis of blood samples from patients with HR-positive/HER2-negative early-stage BC at higher risk of relapse, who have undergone surgery within the previous five years, with no evidence of locoregional, contralateral, or distant disease. Patients must be on adjuvant treatment with ET for at least two years and no more than four years at the time of study enrolment with an additional three years of ET planned. At least 12 months prior to enrolment on the same ET treatment (AI or tamoxifen). For pre-menopausal women and men LHRH is required.

The trial design entails an initial pre-screening phase, a molecular follow-up phase (ctDNA surveillance phase), and an interventional therapeutic phase (treatment phase).

After informed consent is obtained, 1,260 eligible patients will enter a ctDNA surveillance in which primary tumor tissue and matched normal blood will be collected from each patient to obtain a patient-specific somatic mutations panel (tumor signature).

Note: Additional patients may enter the ctDNA surveillance phase if needed, for example if additional arms are opened.

Then, blood will be collected, processed, and analyzed to detect the presence or absence of ctDNA at predefined time points for longitudinal surveillance. ctDNA analysis will occur every three months from study inclusion during the first year and every six months thereafter until positive result or end of accrual.

At the event of ctDNA positivity, patients will be screened to enter the treatment phase of the study. Upon confirmed eligibility, a total of 40 patients will be allocated in one of the following trial's arms adopting a sequential recruitment strategy:

Arm A: Control Arm (N=10) • Patients must continue the same standard ET, prescribed as per standard practice, used in the surveillance phase. Changes in ET are not allowed.

Arm B: Experimental Arm with giredestrant (N=10)

• Giredestrant: 30 mg will be administered PO QD on Days 1 to 28 of each 28-day cycle up to five years or until disease recurrence, unacceptable toxicity, or treatment/study discontinuation (whichever occurs first).

Arm C: Experimental Arm with giredestrant + abemaciclib (N=10)

* Giredestrant: 30 mg will be administered PO QD on Days 1 to 28 of each 28-day cycle up to five years or until disease recurrence, unacceptable toxicity, or treatment/study discontinuation (whichever occurs first).
* Abemaciclib 150 mg will be taken PO BID (two intakes for a total daily dose of 300 mg) during each 28-day cycle up to two years or until disease recurrence, unacceptable toxicity, or treatment/study discontinuation (whichever occurs first).

Arm D: Experimental Arm with giredestrant + inavolisib (N=10)

* Giredestrant: 30 mg will be administered PO QD on Days 1 to 28 of each 28-day cycle up to five years or until disease recurrence, unacceptable toxicity, or treatment/study discontinuation (whichever occurs first).
* Inavolisib: 9 mg will be administered PO QD on Days 1 to 28 of each 28-day cycle up to two years or until disease recurrence, unacceptable toxicity, or treatment/study discontinuation (whichever occurs first).

Note I: In addition to the treatments described on each of the treatment arms, LHRH agonist will be administered to male participants and premenopausal/perimenopausal participants according to local prescribing information. The patient should be supplied with the previous LHRH they were taking.

Note II: During the length of the study, additional treatment arms may open to stay up to date with the most recent advances in oncology, and to be able to provide the best treatment options to patients in this study. Because of that, the N of patients screened to enter the treatment phase may increase.

In the meanwhile, serial assessment of ctDNA will be continuously performed every three months during the first year and every six months thereafter until EoS to correlate any ctDNA variations with response.

Patients discontinuing the study treatment period will enter a post-treatment follow-up period during which survival and new anti-cancer therapy information will be collected every three months (±14 days) from the last dose of study treatment up to the EoS. Telephone contact is acceptable (in some countries medical information can only be shared directly in person with the patient).

Arm extensions

After initiation of study treatments, data obtained from serial assessment of ctDNA will also be used to confirm feasibility of eventual arms extensions, with maximum two arms that could be expanded (10 additional patients will be enrolled in each of the selected arms). The expansion will be approved when the arm complies with the following criteria:

* If at three months, a 90% ctDNA decrease is observed in at least 30% patients and if after three additional months, a 90% ctDNA decrease is maintained in at least 20% patients In this case, 10 additional patients will be enrolled in the specific experimental arms that meet these requirements (N=20).
* If all three experimental arms fulfill the criteria, the two arms with the highest proportion of patients with the highest proportion of 90% decrease will be the ones expanded.
* If cohorts remain too similar (no clear "winners"), the decision will be taken by the Steering Committee based on the duration of the response and the safety and toxicity of each specific treatment.
* If none of the arms fulfill the specific expansion criteria, the Steering Committee will evaluate the data further and may nominate the two arms with the strongest signal of ctDNA decreases for further expansion.

If the strategy of ctDNA monitoring enables physicians to identify patients at high risk of relapse and assess whether treatment at molecular relapse can improve outcome, new cohorts may be added to the study.

ELIGIBILITY:
Inclusion Criteria:

Eligibility criteria for patient registration for ctDNA surveillance phase:

1. Signed informed consent form (ICF) prior to participation in any study-related activities.
2. Male or female patients aged 18 years or older.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
4. Histologically proven primary HR-positive according to the updated American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) 2020 guidelines and HER2-negative BC as per ASCO/CAP 2018 criteria based on local testing on the most recent analyzed biopsy.
5. Patients with high-risk early-stage BC according to at least one of the following criteria:

   1. If no previous neoadjuvant chemotherapy:

   i. pN2/N3 or ii. pN1,

1. pT3/T4 and/or 2. high genomic risk defined as Oncotype Dx Recurrence Score > 25 if post-menopausal; > 20 if pre-menopausal , Prosigna score ≥ 41, Mammaprint high risk category or similar and/or 3. histological grade II/III and Ki67>20%. b. If patients have received previous neoadjuvant chemotherapy, they must have had significant residual invasive disease defined as at least one of the following: i. Residual invasive disease in the breast ypT3 or ypT4. and/or ii. Any macroscopic, ≥ 2 mm, residual lymph node involvement regardless of primary tumor site involvement (includes no residual disease in the breast).

Note: Genomic risk using platforms such as Oncotype Dx, Prosigna or Mammaprint won't be assessed for the screening to participate in the study. However, patients with the detailed scores assessed prior to study inclusion, may be eligible to enter the study if they comply with all the inclusion and exclusion criteria.

6. On adjuvant treatment with ET for at least two years and no more than four years at the time of study enrolment with an additional three years of ET planned. At least 12 months prior to enrolment on the same ET treatment with AI or tamoxifen (luteinizing hormone-releasing hormone [LHRH] for pre-menopausal women and men is required).

Note: Male and pre-menopausal patients treated with tamoxifen alone are excluded.

7. No prior treatment with cyclin-dependent kinases 4/6 (CDK4/6) inhibitors. 8. No prior treatment with fulvestrant. 9. Willingness and ability to provide tissue from one archival tumor tissue sample (either from diagnostic biopsy, primary surgery, or where available from a residual disease post-neoadjuvant therapy).

Note: Patients with multifocal BC may be enrolled, if archival tissue samples from at least two tumors are available and after histopathological examination, all tumors meet pathologic criteria for HR-positive and HER2-negative BC.

10. Absence of metastatic disease by routine clinical assessment (computed tomography [CT] scan of the thorax and abdomen, and bone scan) confirmed no longer than three months prior to study inclusion.

11. Patients must have had surgery for their primary BC with documented clear margins (as per local guidelines) within the past five years.

12. Patients must be able and willing to adhere to study procedures.

Eligibility criteria for entry into the treatment phase:

Patients will be considered eligible to be allocated to standard ET only, giredestrant monotherapy, giredestrant plus abemaciclib, or giredestrant plus inavolisib if they fulfill all the inclusion and none of the exclusion criteria listed below. In order to enter the treatment phase, patients will have had to fulfill first the criteria needed to enter the surveillance phase (which are listed above).

1. Signed ICF prior to study inclusion.
2. ctDNA positivity with no evidence of clinical or radiologic recurrence by standard assessments (e.g.: breast ultrasound, staging scans, RMN).
3. ECOG performance status 0, 1 or 2.
4. Patients must have received the same ET during at least the last 12 months. A temporary discontinuation of < 90 days during the surveillance phase is allowed.
5. Receiving LHRH agonist therapy alongside the same ET treatment for at least 90 days prior to initiation of one of the available study treatments if male or pre-menopausal.
6. Female of reproductive potential and male patients with female partners of childbearing potential, must remain abstinent and truly abstain from sexual activity (refrains from heterosexual intercourse) or use locally recognized adequate methods of contraception (described as that with a failure rate <1%) for the duration of trial treatment. In addition, patients must follow these guidelines for a certain period of time after the last dose of trial treatment, specified in the protocol (Section 7.4.4) depending on which treatment arm the patient is allocated in.

   During this indicated period of time, female and male patients must as well refrain from donating eggs or sperm.

   Note: Female patients will be deemed not of childbearing potential if they are post-menopausal or have had irreversible sterilization. Well-defined pre-menopausal status refers to women who have not reached the post-menopausal state because they are not permanently infertile due to prior bilateral oophorectomy, age ≥60 years or age <60 years with amenorrhea for ≥12 months and estradiol and follicle-stimulating hormone (FSH) levels in the post-menopausal range.
7. Resolution of all acute toxic effects of prior anti-cancer therapy to Grade ≤1 as determined by the National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) version (v) 5.0 (except for alopecia, or other toxicities not considered a safety risk for the patient at investigator's discretion). Adverse events (AEs) of current ET treatment are not included.
8. Adequate hematologic and organ function within 14 days before the first study treatment on Day 1 of Cycle 1, defined by the following:

   • Hematological (without platelet, red blood cell (RBC) transfusion, and/or granulocyte colony-stimulating factor support within 7 days before first study treatment dose): White blood cell (WBC) count > 3.0 x 109/L, absolute neutrophil count (ANC) ≥ 1.5 x 109/L, platelet count ≥ 100.0 x109/L, and hemoglobin ≥ 9.0 g/dL (≥ 5.6 mmol/L).
   * Hepatic: Serum albumin ≥ 3 g/dL; Bilirubin ≤ 1.5 times the upper limit of normal (ULN) (≤ 3 x ULN in the case of Gilbert's disease); aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 × ULN; alkaline phosphatase (ALP) ≤ 2 × ULN.
   * Renal: serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 50 mL/min based on Cockcroft-Gault glomerular filtration rate estimation.
9. Participants who are able and willing to swallow, retain, and absorb oral medication.

Additional inclusion criteria for Arm C (giredestrant + abemaciclib arm)

1. Patients with prior diagnosis of thrombosis might be included as long as they are under stable anti-coagulation regimen therapy 28 days prior to starting treatment with abemaciclib.

Additional inclusion criteria for Arm D (giredestrant + inavolisib arm)

1. Confirmation of biomarker eligibility (detection of specified mutation(s) of PIK3CA via specified test).
2. No prior treatment with any phosphatidylinositol 3-kinase (PI3K), Akt, or mammalian target of rapamycin (mTOR) inhibitors, or any agent whose mechanism of action is to inhibit the PI3K/Akt/mTOR pathway.

Exclusion Criteria for patient registration for ctDNA surveillance phase:

1. Any concurrent or planned treatment for the current diagnosis of BC other than adjuvant ET.
2. Diagnosis of an alternative cancer in the five years prior to primary BC diagnosis other than for non-melanoma carcinoma of the skin or cervical carcinoma in situ. Other stage I tumors will be discussed case by case prior to inclusion with theMedical Monitor of the study. 3.Active or prior documented inflammatory bowel disease (i.e.Crohn's disease, ulcerative colitis, or a preexisting chronic condition resulting in baseline grade ≥1 diarrhea)that may significantly alter the absorption of oral drugs.

4.Active cardiac disease or history of cardiac dysfunction including any of the following:a.History (within two years from screening) or presence of idiopathic bradycardia or resting heart rate <50 beats per minute at screening.b.History of angina pectoris or symptomatic coronary heart disease within 12 months prior to study entry.c.QT interval corrected through use of Fridericia's formula (QTcF) > 450 ms for women and > 470 ms for men by at least three electrocardiograms(ECGs)> 30 minutes apart.d.History or presence of an abnormal ECG that is clinically significant in the investigator's opinion,e.History of ventricular dysrhythmias or risk factors for ventricular dysrhythmias such as structural heart disease (e.g., severe left ventricular systolic dysfunction, left ventricular hypertrophy cardiomyopathy, infiltrative cardiomyopathy, moderate-to-severe valve disease), coronary heart disease (symptomatic or with ischemia demonstrated by diagnostic testing), clinically significant electrolyte EudraCT#: 2022-002616-24Study Code#: MEDOPP485_MIRADORCSP Version 1.0, Date: 23-Dec-202210abnormalities (e.g., hypokalemia, hypomagnesemia, hypocalcemia), or family history of long QT syndrome within 12 months.

5.History of pneumonitis, interstitial lung disease(ILD), or pulmonary fibrosis.

6.Known history of Human Immunodeficiency Virus (HIV) infection(testing not required as part of study screening).

7.Clinically significant liver disease consistent with Child-Pugh C, including active hepatitis (e.g., hepatitis B virus [HBV] or hepatitis C virus [HCV]), current alcohol abuse, cirrhosis, or positive test for viral hepatitis 8.Active bleeding diathesis venous thromboembolism, previous history of bleeding diathesis, or chronic anti-coagulation treatment, or any indications or history of Disseminated Intravascular Coagulation (DIC) or Deep vein thrombosis (DVT). Low molecular weight heparin (LMWH), low dose aspirin or clopidogrel are permitted.

9.Creatinine clearance < 30mL/min. 10.Participants with renal dysfunction who require dialysis. 11.Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the Investigator' opinion cause unacceptable safety risks, contraindicate patient participation in the clinical trial or compromise compliance with the protocol.

12.Females who are known to be breastfeeding or pregnant as determined by a serum pregnancy test,Human chorionic gonadotropin(β-HCG),prior to the administration of any trial treatment. Since β-HCG over expression can be also elevated in some tumor types, a positive result should be confirmed with a validated alternative test (e.g., ultrasound).

13.Female or male participants planning a pregnancy.

Exclusion criteria for entry into the treatment phase:

1. Known hypersensitivity reaction to any investigational or therapeutic compound or their incorporated substances.
2. Undergoing any other simultaneous anti-cancer treatment since enrolling in the study, other than hormonal therapy or a bisphosphonate (or denosumab).
3. Major surgery (defined as requiring general anesthesia) or significant traumatic injury within 28 days of start of study drug, or patients who have not recovered from the side effects of any major surgery.
4. Treatment with strong Cytochrome P450 3A4 (CYP3A4) inhibitors or strong CYP3A4 inducers within 14 days or five drug-elimination half-lives, whichever is longer, prior to initiation of one of the available study treatments.
5. Patient has a history of non-compliance to medical regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1260 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of decrease or clearance in baseline ctDNA at three months after initiation of study treatment | Surveillance phase (up to two years)
  To evaluate the efficacy -in terms of rate of patients with a 90% decrease or clearance in baseline ctDNA at three months- of the different arms.

SECONDARY OUTCOMES:
Total ctDNA detection and breakdown by incidence at first ctDNA test versus incidence at subsequent ctDNA tests. | Surveillance phase (up to two years)
  To assess the incidence of ctDNA detection in patients with HR-positive/HER2-negative BC.
Proportion of patients with at least a 90% decrease in baseline ctDNA at six, nine, and 12 months after initiation of study treatment. | Treatment phase (up to five years)
  To evaluate the efficacy -in terms of a 90% decrease in baseline ctDNA at six, nine, and 12 months- of the experimental arms.
Proportion of patients with at least a 90% decrease in baseline ctDNA at three months maintained at six months and 12 months after initiation of study treatment. | Treatment phase (up to five years)
  To evaluate the efficacy -in terms of a 90% decrease in baseline ctDNA at three months and maintained at six months and 12 months- of the different arms.
Proportion of patients with 50% and 70% decrease in baseline ctDNA at three, six, nine, and 12 months after initiation of study treatment. | Treatment phase (up to five years)
  To evaluate the efficacy -in terms of a 50% and 70% decrease in baseline ctDNA at three, six, nine, and 12 months- of the different arms.
Time to rising ctDNA defined as time to first ctDNA increase compared to baseline | Treatment phase (up to five years)
  To evaluate the efficacy -in terms of time to rising ctDNA during the study follow-up- of the different arms.
Duration of at least a 90% decrease in baseline ctDNA after initiation of study treatment. | Treatment phase (up to five years)
  To evaluate the duration of efficacy -in terms of time with at least a 90% decrease in baseline ctDNA- of the different arms.
Best percentage of ctDNA decrease relative to baseline at six, nine, and 12 months after initiation of study treatment. | Treatment phase (up to five years)
  To evaluate the ctDNA decrease relative to baseline -at three, six, nine, and 12 months- of the different arms.
Number of participants with treatment-related adverse events as assessed by NCI-CTCAE v5.0. | Treatment phase (up to five years)
  National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 will performed to evaluate the safety and tolerability of the different treatments. The occurrence and maximum grade of AEs observed throughout the study will be listed and tabulated according to type and dose level. Any AEs that the investigator reports as unrelated to the drug will also be reported. In this study, side effects will be assessed according to the NCI-CTCAE v.5.0.

OTHER OUTCOMES:
Exploratory endpoint: Time from initiation of study treatment to invasive local/regional recurrence (including ipsilateral invasive breast recurrence) . | Surveillance (up to two years) and treatment (up to five years) phases.
  RFS: Time from initiation of study treatment to invasive local/regional recurrence (including ipsilateral invasive breast recurrence) or distant recurrence or death from any cause. Patients with second primary invasive cancers (breast or non-breast) would be censored at time of detection.
Exploratory endpoint: Genetic studies using tissue and blood samples to investigate the potential association with clinical outcomes, safety, and tolerability profile. | Surveillance (up to two years) and treatment (up to five years) phases.
  Mutation profiling, copy number variability, gene expression, multiplex assays, immunohistochemistry or functional analyses may be performed on tissue, and blood, samples to investigate the potential association with clinical outcomes, safety, and tolerability profile.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Llombart, MD, Principal Investigator — Arnau de Vilanova Hospital, Valencia (Spain)
Locations (32):
- Spain (30):
  - Complejo Hospitalario Universitario A Coruña (CHUAC), A Coruña
  - Hospital General Universitario Dr. Balmis, Alicante
  - Hospital Virgen de los Lirios, Alicante
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital Universitari Dexeus, Barcelona
  - Hospital Universitario de Basurto, Bilbao
  - Hospital Provincial de Castellón, Castellon
  - Hospital Universitario Reina Sofía, Córdoba
  - Institut Català d' Oncologia Girona (ICO), Girona
  - Hospital Universitario Clínico San Cecilio de Granada, Granada
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital Universitario Arnau de Vilanova de Lleida, Lleida
  - Clínica Universidad de Navarra, Madrid
  - Hospital Beata María Ana, Madrid
  - Hospital Universitario de Torrejón, Madrid
  - Hospital Universitario Doce de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Hospitalario Universitario de Navarra, Pamplona
  - Hospital de Sagunto, Sagunto
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitari Sant Joan de Reus, Tarragona
  - Hospital Arnau de Vilanova de Valencia, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia
  - Hospital Universitario La Ribera, Alzira, Valencia
  - Complejo Hospitalario Universitario de Vigo, Vigo
  - Hospital de Xativa, Xàtiva
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (2):
  - Barts Cancer Institute, London
  - Imperial College Healthcare NHS Trust, London

IPD SHARING:
Plan to Share IPD: No